CLINICAL TRIAL: NCT00549666
Title: A Randomized, Placebo-Controlled, Two-Period, Crossover Study to Evaluate the Effect of Lurasidone HCl on Oral Contraceptive Pharmacokinetics in Healthy Female Subjects
Acronym: OC-DDI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: D1050246
Record Dates: First submitted 2007-10-24; First posted 2007-10-26 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Pharmacokinetics
Keywords: OC DDI; lurasidone; Latuda; schizophenia
MeSH Terms: interventions — Lurasidone Hydrochloride; norgestimate, ethinyl estradiol drug combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lurasidone 40 mg (Experimental)
  Interventions: Drug: Lurasidone 40 mg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo 40 mg
- Ortho Tri-Cyclen (Active Comparator)
  Interventions: Drug: Ortho Tri-Cyclen

INTERVENTIONS:
Drug: Lurasidone 40 mg — Lurasidone 40 mg days 12-21 once daily
  Arms: Lurasidone 40 mg
Drug: Placebo 40 mg — Placebo 40 mg once daily during treatment period
  Arms: Placebo
Drug: Ortho Tri-Cyclen — Ortho Tri-Cyclen during 28-day lead in period
  Arms: Ortho Tri-Cyclen

SUMMARY:
A Phase 1, drug, drug, interaction study between Lurasidone HCl and Ortho-tri cyclen

ELIGIBILITY:
Inclusion Criteria:

* Subject is female between 18 and 40 years of age
* Female subjects of reproductive potential will demonstrate a negative serum β-human chorionic gonadotropin level consistent with the non-gravid state at the screening visit
* Subject agrees to take the triphasic oral contraceptive, Ortho Tri-Cyclen™, throughout the study.
* Subject has a history of regular menstrual periods with no substantial breakthrough bleeding episodes while taking Ortho Tri-Cyclen™.
* Subject has a body mass index that is < 33 kg/m2 (see Appendix 1).
* Subject is judged to be in good health
* Subject must have a negative hepatiti and HIV antibody at screening.
* Subject has no clinically significant abnormality on screening ECG.

Exclusion Criteria:

* Subject has a history of major GI abnormalities/peptic ulceration, hematological, genitourinary, cardiovascular (including hypertension), renal, hepatic, pulmonary, psychiatric, endocrine (including diabetes) or metabolic (including glaucoma), neurologic or cerebrovascular disease, or any history of cancer.
* Subject has systolic blood pressure ≥ 140 mm Hg and/or diastolic blood pressure ≥ 90 mm Hg at screening.
* Subject has a history of any chronic and/or active hepatic disease including elevations of serum transaminases, hepatitis, biliary tract disease, or a history of any gastrointestinal surgery.
* Subject has any other acute or chronic medical or psychiatric condition that, in the opinion of the investigator, would limit the patient safety or confound the results of the study.
* Subject has an ECG at screening with PR > 240 msec; QRS complex > 120 msec; QTcB > 450; or any significant morphologic changes other than nonspecific T-wave changes.
* Subject is currently a user of any illicit drugs (including "recreational use") including marijuana, or has recently used illicit drugs, or has a history of drug or alcohol dependence in the past year or abuse within the last 3 months.
* Subject consumes excessive amounts of alcohol
* Subject has had surgery within last 12 weeks, donated a unit of blood (within 4 weeks), or participated in another clinical study within 30 days of screening.
* Subjects with hypertension, hyperlipidemia, and diabetes should also be excluded. (See package circular under "Contraindications")
* Subject has clinically significant abnormalities at screening clinical examination or laboratory safety tests
* Subject has a prolactin level of over 200 ng/mL at screening.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2007-08; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (1):
- Covance Global Clinical Pharmacology, Inc., San Diego, California, United States